



IRAS ID: 242462

## **Informed Consent Form**

## Assessing gut permeability using spectroscopy

Study title: Non-invasive transcutaneous spectroscopy for the assessment of gut permeability (GutPerm)

IRAS Project ID: 242462

| Pat | tient Trial ID Number: | |
|---|---|---|
| Na | me of Principal Investigator: <u>Dr Alex Thompson</u> | |
| Name of patient to whom this ICF applies: | | |
| | Please | e initial boxes |
| 1. | I confirm that I have read and understand the Participant Information Sheet "Assessing gut permeability using spectroscopy v4.2A 01-May-2019" for the above study and have had the opportunity to ask questions about the study and understand what is involved. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or other legal rights being affected, and I understand that any remaining samples will be destroyed at my request, but data collected up to the point of my withdrawal may still be used. | |
| 3. | I agree to have a 'Spectroscopic gut permeability test' and understand that there is a small risk of nausea and other allergic reactions (including anaphylaxis) with this test. | |
| 4. | I agree to provide two 5 ml blood samples during my study visit (equivalent to approximately one teaspoon of blood for each sample). | |
| | If you do <u>NOT</u> consent to provide two 5 ml blood samples, please put a line through all of point 4 above, and do <u>NOT</u> initial the box as indicated – you can still participate in the main trial. | |
| 5. | I agree to provide two urine samples during my study visit. | |
| | If you do $\underline{NOT}$ consent to provide two urine samples, please put a line through all of point 5 above, and do $\underline{NOT}$ initial the box as indicated – you can still participate in the main trial. | |
| 6. | I agree to provide one or more stool samples within approximately 48 hours of my study visit. | |
| | If you do $\underline{NOT}$ consent to collection of a stool sample, please put a line through all of point 6 above, and do $\underline{NOT}$ initial the box as indicated – you can still participate in the main trial. | |
| 7. | I agree to have a 'PEG permeability test' and understand that there is a small risk of diarrhoea and bloating with this test. | |
| 8. | I agree to allow information about me to be collected, analysed, reported and transferred to other approved collaborators within and outside the European Economic Area for healthcare and/or medical research purposes. I understand that my identity will remain anonymous. | |
| 9. | I give consent for any of the blood, urine and stool samples that I give that are used as part of this study to be used in future research projects that comply with regulations and which have approval from an independent research ethics committee. This may include transfer of my samples outside | |





IRAS ID: 242462

of the European Economic Area. Under these circumstances my samples will be retained for up to 10 years in Imperial College's secure and fully regulated Biobank.

If you do  $\underline{NOT}$  consent to your samples being stored and used for future research in this way, please put a line through all of point 9 above, and do  $\underline{NOT}$  initial the box as indicated – you can still participate in the main trial.

| | still participate in the main trial. | | , |
|---|---|---|---|
| 10. | I agree to have a second 'Spectr' hyperosmotic' solution. I understand with the 'Spectroscopic gut pern' hyperosmotic solution' is minimal. | d that there is a small risk of nau | usea or other allergic reactions |
| | If you do <u>NOT</u> consent to have a sebeen approached about this section and do <u>NOT</u> initial the box as indicated | n of the study, please put a line | through all of point 10 above, |
| 11. | I wish to be contacted by e-mail with a summary of the research findings once the study is complete. Your e-mail address will not be used for any other purpose. | | |
| | Contact e-mail: | | |
| If you do <u>NOT</u> wish to be contacted regarding the study results, please put a line through all of point 11 above, do <u>NOT</u> leave a contact e-mail address and do <u>NOT</u> initial the box as indicated – you can still participate in the main trial. | | | |
| 12. I agree to take part in the study. | | | |
| Ple | ase sign and date below. | | |
| Naı | me of Subject | Signature | Date |
| Naı | me of Person taking consent | <br>Signature | <br>Date |

1 copy for subject; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes